CLINICAL TRIAL: NCT00792350
Title: International Study With Nexavar About Safety and Efficacy in Carcinoma Hepatocellular Therapy (HCC)
Brief Title: INSIGHT - Post Marketing Surveillance
Acronym: INSIGHT
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 14690; 13419 (Other: Company internal); 13420 (Other: Company internal); NX0801DE (Other: Company internal); NX0801AT (Other: Company internal); NX0801 (Other: Company internal)
Record Dates: First submitted 2008-11-14; First posted 2008-11-17 (Estimated); Last update posted 2014-05-14 (Estimated); Status verified 2014-05

CONDITIONS: Carcinoma, Hepatocellular
Keywords: Carcinoma, Hepatocellular; Sorafenib
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Sorafenib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1
  Interventions: Drug: Sorafenib (Nexavar, BAY43-9006)

INTERVENTIONS:
Drug: Sorafenib (Nexavar, BAY43-9006) — Treatment of Hepatocellular Carcinoma with Nexavar (HCC)

SUMMARY:
In this international non-interventional post-marketing surveillance study we want to evaluate patient characteristics in HCC patients as well as efficacy and safety of Sorafenib (Nexavar®) treatment under daily-life treatment conditions. Specifically investigated are the tumor status, prior and/ or concomitant surgical, radiological and drug treatment and the duration of Sorafenib treatment.

ELIGIBILITY:
Inclusion Criteria:

* In- and outpatients with diagnosis of hepatocellular carcinoma (HCC) and decision taken by the investigator to prescribe Nexavar

Exclusion Criteria:

* Exclusion criteria must be read in conjunction with the local product information

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In and outpatients with diagnosis of hepatocellular carcinoma (HCC) and decision taken by the investigator to prescribe Nexavar.
Sampling Method: Non-Probability Sample
Enrollment: 791 (Actual)
Dates: Start 2008-04; Primary Completion 2013-10 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Efficacy: status of tumor, patients performance status | At each follow-up visit, every 2-4 months

SECONDARY OUTCOMES:
Duration of treatment | At each follow-up visit, every 2-4 months
Time of survival | At each follow-up visit, every 2-4 months
Reports of adverse events | At each follow-up visit, every 2-4 months

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (2):
- Many Locations, Austria
- Many Locations, Germany